CLINICAL TRIAL: NCT01943617
Title: Optimized Treatment and Regression of HBV-induced Compensated Liver Cirrhosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Peking University People's Hospital (Other); RenJi Hospital (Other); Peking University (Other); Shanghai Zhongshan Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Public Health Clinical Center (Other Government); Nanfang Hospital, Southern Medical University (Other); Sir Run Run Shaw Hospital (Other); Beijing YouAn Hospital (Other); Peking University First Hospital (Other); Beijing 302 Hospital (Other); Peking Union Medical College Hospital (Other); Beijing Ditan Hospital (Other); Beijing Tiantan Hospital (Other); Huashan Hospital (Other); Tongji Hospital (Other); Tang-Du Hospital (Other); Fifth Hospital of Shijiazhuang City (Other); Logistics University of Chinese People's Armed Police Forces (Other); The First Affiliated Hospital of Shanxi Medical University (Other); The Affiliated Hospital of Yanbian University (Other)
Responsible Party: Principal Investigator, Hong You, Vice-Director Liver Research Centre, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013ZX10002004-3
Record Dates: First submitted 2013-09-05; First posted 2013-09-17 (Estimated); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Liver Cirrhosis
Keywords: Liver Cirrhosis; Hepatitis B; Compensation; Efficacy
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis B | interventions — entecavir; Thymalfasin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Entecavir Therapy (Active Comparator): Entecavir, 0.5mg, qd, oral, for 2 years
  Interventions: Drug: Entecavir
- Entecavir plus thymosin therapy (Experimental): Entecavir plus thymosin-α 1.6μg, Twice a week, ih, in the middle one year
  Interventions: Drug: Entecavir; Drug: Thymosin-α

INTERVENTIONS:
Drug: Entecavir — anti-viral therapy
  Other Names: Entecavir dispersible tablets
Drug: Thymosin-α — anti-viral and antitherapy
  Other Names: Zadaxin
  Arms: Entecavir plus thymosin therapy

SUMMARY:
Six hundreds patients with chronic hepatitis B clinically diagnosed as compensated liver cirrhosis are randomly assigned in a 1:1 ratio. One arm is entecavir alone for 2 years; the other is entecavir alone for the first 0.5 year, entecavir plus thymosin-α for 1 year, entecavir for another additional 0.5 year.Patients will be assessed at baseline, at every six months for blood cell count, liver function test, HBVDNA, AFP, prothrombin time, liver ultrasonography, and Fibroscan;

ELIGIBILITY:
Inclusion Criteria:

1. Patients from age 18 to 65 years ;
2. Male or female;
3. Treatment-naive patients of clinically diagnosed as HBV-induced compensated cirrhosis(meet one of the following two criterions);

   1. endoscopy: esophageal varices , exclusion of noncirrhotic portal hypertension
   2. if no endoscopy,should meet two of the four Criterias:

      * Imaging (US, CT or MRI, et al) showing Surface nodularity: Echogenecity
      * Platelet (PLT) < 100×10 < 9 >/L , no other interpretation
      * Albumin (ALB) < 35.0 g/L, or International Standard Value (INR) > 1.3 (Prothrombin Time (PT) prolonged > 3s), or Cholinesterase (CHE) decrease
      * Liver stiffness measurement value > 12.4 kpa (ALT<5×ULN)
4. HBeAg-positive, HBVDNA > 2×10<3> IU/ml or with HBeAg-negative patients, HBVDNA > 2×10<2> IU/ml;
5. Agree to be followed up regularly;
6. Signature of written inform consent.

Exclusion Criteria:

1. Patients with decompensated cirrhosis: including ascites, hepatic encephalopathy, esophageal varices bleeding or other complications of decompensated cirrhosis or hepatocelluar carcinoma;
2. Patients who are allergic to entecavir, thymosin or their components, and those considered not suitable for medicine in this study;
3. Patients with HCV or HIV infection, alcoholic liver disease, autoimmune liver disease, genetic liver disease, drug-induced liver injury, severe non-alcoholic fatty liver disease or other chronic liver diseases;
4. Patients with baseline AFP level higher than 100ng/ml and possible malignant lesion on image, or AFP level higher than 100ng/ml for more than three months;
5. Creatinine > 1.5×ULN;
6. Patients with other uncured malignant tumors;
7. Patients with severe diseases of heart, lung, kidney, brain, blood system or other organs;
8. Patients with any other reasons not suitable for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2013-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Decompensated rate of Liver Cirrhosis after 2 years treatment | 2 years
  Decompensated rate of Liver Cirrhosis (ascites, hepatic encephalopathy, esophageal varices bleeding and Hepatocellular Carcinoma) after 2 years treatment.

SECONDARY OUTCOMES:
Child-Pugh and MELD scores | 1 and 2-year
  The progress of Child-Pugh and MELD scores after 1 and 2-year treatment
The HBV DNA undetectable rate | 1 and 2-year
  The HBV DNA undetectable rate after 1 and 2-year treatment
Liver stiffness measurement | 1 and 2-year
  Liver stiffness measurement change after 1 and 2-year treatment.
Quality of Life | 1 and 2-year
  Quality of life after 1 and 2-year treatment by SF-36 and EQ-5D questionares

CONTACTS AND LOCATIONS:
Overall Officials: Hong You, Doctor, Principal Investigator — Beijing Friendship Hospital
Locations (21):
- China (21):
  - Beijing Ditan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - 302 Military Hospital Of China, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing YouAn Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - PeKing University, Beijing, Beijing Municipality
  - NanfangHospital,Southern Medical University, Guangzhou, Guangdong
  - Shijiazhuang Fifth Hospital, Shijiazhuang, Hebei
  - Tongji Hospital, Tongji Medical College ,Huazhong University of Science ＆Technology, Wuhan, Hubei
  - Sir Run Run Shaw Hospital,School of Medicine,Zhejiang University, Hangzhou, Jiangsu
  - The Affiliated Hospital of Yanbian University, Yanbian, Jilin
  - RenjiHospital,Shanghai Jiao Tong University,School of Medicine, Shanghai, Shanghai Municipality
  - Huashan Hospital FuDan University, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - The Hospital Affiliated to Logistics University of Chinese People's Armed Police Force, Tianjin, Tianjin Municipality

REFERENCES:
- [Derived] Wu X, Hong J, Zhou J, Sun Y, Li L, Xie W, Piao H, Xu X, Jiang W, Feng B, Chen Y, Xu M, Cheng J, Meng T, Wang B, Chen S, Kong Y, Ou X, You H, Jia J. Health-related quality of life improves after entecavir treatment in patients with compensated HBV cirrhosis. Hepatol Int. 2021 Dec;15(6):1318-1327. doi: 10.1007/s12072-021-10240-4. Epub 2021 Nov 29. PMID 34843068
- [Derived] Wu X, Zhou J, Sun Y, Ding H, Chen G, Xie W, Piao H, Xu X, Jiang W, Ma H, Ma A, Chen Y, Xu M, Cheng J, Xu Y, Meng T, Wang B, Chen S, Shi Y, Kong Y, Ou X, You H, Jia J. Prediction of liver-related events in patients with compensated HBV-induced cirrhosis receiving antiviral therapy. Hepatol Int. 2021 Feb;15(1):82-92. doi: 10.1007/s12072-020-10114-1. Epub 2021 Jan 18. PMID 33460002